CLINICAL TRIAL: NCT07177521
Title: Primary Stability and Peri-implant Outcomes of Short Implants in Post-extraction Single-tooth Sites: a Randomized Controlled Trial.
Brief Title: Primary Stability and Peri-implant Outcomes of Short Implants in Post-extraction Single-tooth Sites
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Post-extraction-implants
Record Dates: First submitted 2025-09-08; First posted 2025-09-17 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Edentulous Jaw; Tooth Loss; Toothless Mouth
MeSH Terms: conditions — Jaw, Edentulous; Tooth Loss; Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Socket grafting with a fully resorbable synthetic biomaterial (β-tricalcium phosphate + calcium sulfate).
  Interventions: Procedure: Insertion of implants in post-extraction tooth
- Group 2 (Active Comparator): Socket grafting with a xenograft and a custom Sealing Socket Abutment with a concave emergence profile.
  Interventions: Procedure: Insertion of implants in post-extraction tooth

INTERVENTIONS:
Procedure: Insertion of implants in post-extraction tooth — Two widely used approaches include:
  1. Socket grafting with a fully resorbable synthetic biomaterial (β-tricalcium phosphate + calcium sulfate).
  2. Socket grafting with a xenograft and a custom Sealing Socket Abutment (SSA) with a concave emergence profile.
  No randomized controlled trials have yet compared these protocols with integrated outcomes including resonance frequency analysis, peri-implant health indices, radiographic bone level changes, and digital intraoral scanning (IOS)-based morphometric analysis.

SUMMARY:
The placement of short implants in post-extraction sockets is a valuable option when residual bone height is limited, minimizing morbidity and treatment time. The management of the peri-implant gap and soft tissues may influence primary stability, hard/soft tissue remodeling, and implant success.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Single-tooth post-extraction sites requiring immediate implant placement in posterior regions (premolars/molars) or selected anterior sites.
* Planned short implant (≤7-8 mm length, 3.5-5.0 mm diameter).
* Adequate oral hygiene, no active periodontal disease.
* Written informed consent.

Exclusion Criteria:

* Heavy smoking (>20 cigarettes/day).

  * Uncontrolled diabetes or systemic conditions affecting bone healing.
  * Current bisphosphonate/antiresorptive therapy.
  * Immunosuppression, pregnancy.
  * Poor oral hygiene or acute infection at site.
  * Severe bone dehiscence preventing primary stability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Primary stability | 1 month
  To compare the primary stability (ISQ values at implant insertion) of short implants placed in post-extraction sockets using the two grafting protocols.

SECONDARY OUTCOMES:
Clinical Indices | 12 months
  To assess peri-implant health indices (PD)
Clinical Indices | 12 month
  To assess peri-implant health indices (BoP)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe D'Albis, Dr, Principal Investigator — University of Bari Aldo Moro; Saverio Capodiferro, Prof, Study Chair — University of Bari Aldo Moro
Locations (1):
- University of Bari Aldo Moro, Bari, Italy

IPD SHARING:
Plan to Share IPD: No